CLINICAL TRIAL: NCT03336710
Title: Decentering in Daily Life: Underlying Mechanisms and Impact on Well-Being
Brief Title: Perspective on Thoughts and Feelings as a Predictor of Psychological Well-being in Daily Life, in a Community Sample
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Kenneth G. DeMarree, Assistant Professor of Psychology, State University of New York at Buffalo
Other Study IDs: 1R21AT009470-01 (NIH); R21AT009470 (NIH)
Record Dates: First submitted 2017-10-25; First posted 2017-11-08 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Mental Health; Mindfulness
Keywords: Self-control; Ecological Momentary Assessment; Attentional bias; Respiratory Sinus Arrhythmia; Affect; Emotion Regulation; Well-being; Decentering; Affective disorders
MeSH Terms: conditions — Psychological Well-Being; Self-Control; Arrhythmia, Sinus; Emotional Regulation; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary sample: Community sample of adults (18-65) from the greater Buffalo, NY region, oversampling people who are seeking mental health treatment.

SUMMARY:
This project examines the psychological construct of decentering - a mindfulness-related construct marked by an observer perspective on one's ongoing mental processes. Specifically, this project seeks to explore the extent to which decentering modulates the relationship between people's affective states and their momentary mental health and well-being, and to test the psychological processes by which decentering might exert these effects. This study includes a baseline assessment followed by a 7-day study completed from home where participants respond to brief surveys about their current experiences six times per day (i.e., an Ecological Momentary Assessment [EMA] design).

The investigators hypothesize that decentering moderates the association of extreme affect with related symptoms (i.e., elevated negative affect with depression and anxiety; elevated positive affect with mania, narcissism, and histrionic traits) and well-being, such that the association is attenuated at high levels of decentering. This will be examined using the EMA data, analyzing between-person levels (i.e., trait) as well as momentary within-person processes (i.e., concurrent and prospective states).

Further, the investigators predict that broadened attentional focus and improved self-regulation are mechanisms that contribute to the beneficial effects of decentering in daily life. This hypothesis will be examined in two ways:

1. as individual differences, wherein greater self-regulatory abilities (e.g., higher heart rate variability) and less attentional biases towards emotional stimuli mediate the association between trait decentering and subsequent daily well-being/symptoms, and
2. as within-person momentary levels, wherein broader attentional processes and greater self-regulation in daily life mediate the concurrent and prospective association between momentary decentering and well-being/symptoms.

Note that the study uses a multimodal assessment of each of the proposed processes. For attentional processes, a variety of parameters extracted from an emotional eye tracking paradigm will be examined. For self-regulatory abilities, assessments will include self-report, physiological (heart rate variability), and behavioral ("go / no-go" task) measures of such abilities.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65, fluency in English

Exclusion Criteria:

* current cognitive impairments (i.e., intellectual disability, dementia, current psychotic symptoms) that preclude giving informed consent and accurately answering study questions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population from which the sample will be recruited will be residents of the greater Buffalo, NY metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Momentary psychological distress | 6 x daily for 7 days following the baseline assessment
  2 items (developed new for this study) assessing the presence and impact of idiographic symptoms identified at baseline, and 4 items assessing dysphoria adapted from the Inventory of Depression and Anxiety Symptoms (IDAS)
Momentary eudaimonic well-being | 6 x daily for 7 days following the baseline assessment
  2 items assessing eudaimonic well-being adapted from Breines et al. (2008) and Lambert et al. (2013)
Momentary hedonic well-being (state positive and negative affect) | 6 x daily for 7 days following the baseline assessment
  8 items assessing hedonic well-being (positive and negative affect), taken from the Positive and Negative Affect Schedule (PANAS).
State Decentering | 6 x daily for 7 days following the baseline assessment
  4 items assessing current decentering, adapted from Fresco et al. (2007), Gillanders et al. (2014), and Shoham et al. (2017)
Trait Decentering: Experiences Questionnaire | Baseline session only
  Experiences Questionnaire is a trait measure of decentering, which assesses the Observer Perspective aspect of decentering. From Fresco et al., (2007)
Trait decentering: Valence free decentering measure | Baseline session only
  This is an in-development measure of decentering that measures the construct of decentering without explicitly referring to negative thoughts and feelings.
Trait decentering: Cognitive Fusion Questionnaire | Baseline session only
  The Cognitive Fusion Questionnaire is a decentering measure that assesses the Reduced Struggle with Inner Experiences aspect of decentering. From Gillanders et al., (2014).
Trait decentering: Toronto Mindfulness Scale-Decentering Subscale | Baseline session only
  The Toronto Mindfulness Scale-Decentering subscale is a decentering measure that assesses the Observer Perspective aspect of decentering. From Davis, Lau, & Cairns (2009).

SECONDARY OUTCOMES:
Self-reported momentary self-regulation | 6 x daily for 7 days following the baseline assessment
  3 questions assessing current perceived willpower & mental exhaustion, adapted from Davisson (2013) and Milyavskaya & Inzlicht (2017).
Self-reported momentary attentional focus | 6 x daily for 7 days following the baseline assessment
  4 attentional emotion regulation items (distraction, positive rumination, negative rumination, and reappraisal) adapted from Brans et al. (2013), Feldman et al. (2008), and Nolen-Hoeksema & Morrow (1991)
Baseline self-regulation: Go/no-go task | Baseline session only
  Go/no-go task asks people to respond to a large number of "go" trials (80%) and a smaller number of "no go" trials. The ability to inhibit the dominant "go" response is seen as an operative measure of self-regulatory abilities, consequently the number of "no go" signals responded to is one measure of self-regulatory abilities.
Baseline self-regulation: Resting heart rate variability | Baseline session only
  Assessed with a Polar V800 athletic watch during a 5-minute vanilla baseline and a 5-minute paced breathing task.
Baseline self-regulation: Self-Control Scale (short form) | Baseline session only
  A self-report measure of people's perceived self-control abilities and outcomes, developed by Tangney, Baumeister, & Boone (2004).
Baseline attentional breadth: Emotional eye-tracking paradigm | Baseline session only
  Participants will view a series of emotionally expressive versus neutral faces, and the fixation time and number of fixations towards emotionally evocative (angry, sad, happy) faces will serve as indicators of attentional bias
Baseline attentional breadth: Thought Control Questionnaire | Baseline session only
  Self-report measure corresponding to various emotion regulation strategies (distraction and reappriasal)
Baseline attentional breadth: Responses to Positive Affect Scale | Baseline session only
  Self-report measure corresponding to various emotion regulation strategies (positive rumination)
Baseline attentional breadth: Ruminative Responses Scale | Baseline session only
  Self-report measure corresponding to various emotion regulation strategies (negative rumination)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Gainey, Ph.D., Principal Investigator — University at Buffalo; Kenneth G DeMarree, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Department of psychology, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Materials will be made available 6 months after publication of the primary outcomes.
Access Criteria: Data and study materials relevant to any publication will be posted within 6 months of publication on the open science framework, which will be accessible by any interested party.

REFERENCES:
- [Background] Naragon-Gainey K, DeMarree KG. Structure and validity of measures of decentering and defusion. Psychol Assess. 2017 Jul;29(7):935-954. doi: 10.1037/pas0000405. Epub 2016 Oct 31. PMID 27797554
- [Background] Bernstein A, Hadash Y, Lichtash Y, Tanay G, Shepherd K, Fresco DM. Decentering and Related Constructs: A Critical Review and Metacognitive Processes Model. Perspect Psychol Sci. 2015 Sep;10(5):599-617. doi: 10.1177/1745691615594577. PMID 26385999
- [Background] Shoham A, Goldstein P, Oren R, Spivak D, Bernstein A. Decentering in the process of cultivating mindfulness: An experience-sampling study in time and context. J Consult Clin Psychol. 2017 Feb;85(2):123-134. doi: 10.1037/ccp0000154. PMID 28134540
- [Background] Naragon-Gainey K, DeMarree KG. Decentering attentuates the associations of negative affect and positive affect with psychopathology. Clinical Psychological Science. Epub 2017 Aug 11.
- [Background] Tangney JP, Baumeister RF, Boone AL. High self-control predicts good adjustment, less pathology, better grades, and interpersonal success. J Pers. 2004 Apr;72(2):271-324. doi: 10.1111/j.0022-3506.2004.00263.x. PMID 15016066
- [Background] Fresco DM, Moore MT, van Dulmen MH, Segal ZV, Ma SH, Teasdale JD, Williams JM. Initial psychometric properties of the experiences questionnaire: validation of a self-report measure of decentering. Behav Ther. 2007 Sep;38(3):234-46. doi: 10.1016/j.beth.2006.08.003. Epub 2007 Apr 24. PMID 17697849
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Watson D, O'Hara MW, Simms LJ, Kotov R, Chmielewski M, McDade-Montez EA, Gamez W, Stuart S. Development and validation of the Inventory of Depression and Anxiety Symptoms (IDAS). Psychol Assess. 2007 Sep;19(3):253-68. doi: 10.1037/1040-3590.19.3.253. PMID 17845118
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575